CLINICAL TRIAL: NCT05833932
Title: Suhexiang Pill for Acute Ischemic Stroke: A Prospective Registry Study of Real-world Data
Brief Title: Suhexiang Pill for Acute Ischemic Stroke: A Registry Study
Acronym: SUNRISE
Status: Recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Other Study IDs: 2021XS-001-05
Record Dates: First submitted 2023-03-24; First posted 2023-04-27 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; traditional Chinese medicine; registry study
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Suhexiang Pill — Suhexiang Pill is an approved traditional Chinese patent medicine.

SUMMARY:
The primary purpose of this study is to investigate the effectiveness and safety of the Suhexiang Pill for patients with acute ischemic stroke in real-world settings.

DETAILED DESCRIPTION:
Suhexiang Pill, a traditional Chinese patent medicine, is widely used in China for acute stroke. However, there is a lack of evidence of its efficacy and safety for acute ischemic stroke in real-world setting. This registry study will recruit 1000 patients who receive Suhexiang Pill treatment after acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke within 7 days of symptom onset.
* Age ≥ 18
* Patient who has received Suhexiang Pill treatment
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Be allergic to Suhexiang Pill
* Known to be pregnant or breastfeeding.
* With conditions that render outcomes or follow-up unlikely to be assessed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Acute ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients independent | 90 days
  Proportion of patients independent is defined as the modified Rankin Scale score of 0, 1, or 2.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale | The change from baseline to day 10 or discharge.
  The National Institute of Health Stroke Scale (NIHSS) ranges from 0 to 42, with higher scores indicating more severe neurological deficits.
Glasgow Coma Scale | The change from baseline to day 10 or discharge.
  The Glasgow Coma Scale (GCS) is used to describe the extent of impaired consciousness in all types of acute medical and trauma patients, ranging from 0 to 15, with lower scores indicating more severe impaired consciousness.
Patient reported outcome | At day 10 or discharge.
  The patient reported outcome (PRO) scale of stroke consists of four dimensions including the influence on physical, emotional, and social functioning, as well as the overall satisfaction with treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lai X, Xiong X, Jia Q, Liu T, Yang Z, Zhang C, Kong L, Cao K, Dong T, Fang C, Ge J, Dong L, Zong Z, Chen S, Ma Y, Bai X, Wu D, Xie Y, Zhang M, Wang Y, Jiang G, Song D, Wang Y, Gui C, Geng Q, Gao Y; SUNRISE study investigators. Suhexiang pill for acute ischemic stroke in real-world practice setting (SUNRISE): protocol of a multicenter registry. BMC Complement Med Ther. 2025 Jan 28;25(1):30. doi: 10.1186/s12906-025-04762-9. PMID 39875901